CLINICAL TRIAL: NCT04437589
Title: Opioid-Free Intravenous Anesthesia for Patients With Joint Hypermobility Syndrome Undergoing Craneo-Cervical Fixation: A Case-series Study Focused on Anti-hyperalgesic Approach
Brief Title: Opioid-Free Anesthesia for Patients With Joint Hypermobility Syndrome Undergoing Craneo-Cervical Fixation: A Case-series
Status: Completed | Type: Observational
Sponsor: Servei Central d'Anestesiologia (Other)
Responsible Party: Principal Investigator, Carlos Ramirez Paesano, Principal Investigator, Servei Central d'Anestesiologia
Other Study IDs: OPIOIDANALGESIA1
Record Dates: First submitted 2020-06-11; First posted 2020-06-18 (Actual); Last update posted 2020-07-10 (Actual); Status verified 2020-07

CONDITIONS: Ehlers-Danlos Syndrome; Craniocervical Syndrome
Keywords: Craneocervical -instability; Craneocervical -fixation; Opioid induced hyperalgesia; Free-opioid-anesthesia; Ehlers-Danlos Syndrome; Joint Hipermobility syndrome; Central sensitization phenomena
MeSH Terms: conditions — Ehlers-Danlos Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Exposure group: In this group the treatment applied for postoperative pain involves Free-opioid anesthesia (LKDi).
- Control group: In this group the treatment applied for postoperative pain involves an opioid-based anesthesia.

SUMMARY:
Cranio-cervical instability (CCI) has been well identified in diseases regarding connective tissue, such as Ehlers-Danlos Syndrome/Hipermobility Type (EDS-HT). These patients frequently suffer from severe widespread pain with very difficult management and control. Chronic neuroinflamation, opioid-induced hyperalgesia, and central sensitization phenomena may explain this complex painful condition. A retrospective, observational, consecutive case series study is designed to determine if opioid-free anesthetic management shows a reduction in postoperative pain and opioid rescues needs in comparison with opioid-based anesthesia management for patients with EDS-HT undergoing crano-cervical fixation.

DETAILED DESCRIPTION:
Cranio-cervical instability (CCI) has been well identified in diseases regarding connective tissue, such as Ehlers-Danlos Syndrome/Hipermobility Type (EDS-HT). These patients frequently suffer from severe widespread pain with very difficult management and control. Chronic neuroinflamation, opioid-induced hyperalgesia, and central sensitization phenomena may explain this complex painful condition. A retrospective, observational, consecutive case series study is designed to determine if opioid-free anesthetic management shows a reduction in postoperative pain and opioid rescues needs in comparison with opioid-based anesthesia management for patients with EDS-HT undergoing craneo-cervical fixation.

Main Aim: To determine if the administration of opioid-free anesthesia with propofol, lidocaine, ketamine, and dexmedetomidine shows reduction of postoperative pain, and postoperative needs of opioids rescue in patients undergoing CCF.

Secondary Aims:

* To determine if the administration of opioid-free anesthesia in patients undergoing CCF, and postoperative Lidocaine, Ketamine, and Dexmedetomidine infusions can reduce the preoperative needs of opioids treatment at discharge time.
* To determine if the administration of opioid-free anesthesia in patients undergoing CCF reduces the postoperative gastrointestinal complications.
* To determine if the administration of postoperative Lidocaine, Ketamine, and Dexmedetomidine infusions in patients underwent CCF can reduce the preoperative needs of postoperative anxiolytic treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of Hypermobility Syndrome undergoing Craneo-cervical fixation (CCF)
* Patients between 18-60 years.
* Patients enrolled in CCF surgery between September 2018 to March 2020 to get stabilized craneo-cervical instability (CCI).
* Patients under opioid-based total intravenous anesthesia or opioid-free total intravenous anesthesia with lidocaine, ketamine and dexmedetomidine (LKD).

Exclusion Criteria:

* CCF to stabilized post-traumatic or oncologic CCI.
* Lidocaine allergy.
* Advances heart-block.
* Epilepsy or convulsive syndrome non-medicated.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients between 18-60 years with diagnosis of Hypermobility Syndrome undergoing Craneo-cervical fixation (CCF) between Sept, 2018 to March, 2020 to get stabilized craneo-cervical instability (CCI), and performed under opioid-based total intravenous anesthesia or opioid-free total intravenous anesthesia with lidocaine, ketamine and dexmedetomidine (LKD).
Sampling Method: Non-Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2018-09-06 (Actual); Primary Completion 2020-03-09 (Actual); Study Completion 2020-03-09 (Actual)

PRIMARY OUTCOMES:
Age | Baseline
  Patient's age when the surgery was performed (in years)
Sex | Baseline
  Patient sex classified in two groups: female (1) and male (2)
PO Analgesia | Baseline
  Postoperative analgesia is a nominal variable which indicates the type of analgesia administered to the patient.
  There are 4 options: Lidocaine-Ketamine-Dexmetodimine (LKDi) as group 1, PCA morphine infusion pump as group 2, Ketamine perfusion as group 3 and Methadone-Ketamine as group 4.
Preoperative EVA | Baseline
  Escala Visual Analógica de dolor (EVA) is an analogic visual scale to measure the patients pain. It has a range between 0 and 10. Higher values mean more pain.
  The Preoperative EVA measures the pain before the surgery. If there is more than one measure the result is presented as the mean of all measurements.
Preoperative Opioids | Baseline
  The preoperative opioids is a categorical variable that indicates if the patient took opioids before the surgery.
  There are 4 options:
  * No opioids or eventually taken as option 0
  * Weak opioids (tramadol, codeine, trapentadol) as option 1
  * Strong opioids (fentanile, oxicodone, morphine, buprenorphine) as option 2
  * A combination of strong opioids as option 3
Postoperative EVA 1 | 1 day after surgery
  Escala Visual Analógica de dolor (EVA) is an analogic visual scale to measure the patients pain. It has a range between 0 and 10. Higher values mean more pain.
  The postoperative EVA 1 is measured 1 day after surgery.
Postoperative EVA 2 | 2 days after surgery
  Escala Visual Analógica de dolor (EVA) is an analogic visual scale to measure the patients pain. It has a range between 0 and 10. Higher values mean more pain.
  The postoperative EVA 2 is measured 2 day after surgery.
Postoperative EVA 4 | 4 days after surgery
  Escala Visual Analógica de dolor (EVA) is an analogic visual scale to measure the patients pain. It has a range between 0 and 10. Higher values mean more pain.
  The postoperative EVA 4 is measured 4 day after surgery.
Postoperative EVA 6 | 6 days after surgery
  Escala Visual Analógica de dolor (EVA) is an analogic visual scale to measure the patients pain. It has a range between 0 and 10. Higher values mean more pain.
  The postoperative EVA 6 is measured 6 day after surgery.
Sufentanil doses 1 | From surgery release till first day of hospitalization
  Number of pills of sufentanil that the patient has token besides the main treatment. The variable is gathered 1 day after surgery.
  Sufentanil doses 1 is a categorical variable with 4 levels:
  * From 0 to 2 pills (equal or less than 30mcg/day) as level 1.
  * From 2 to 4 pills (from 30mcg/day to 60mcg/day)
  * From 5 to 10 pills (from 75mcg/day to 150 mcg/day)
  * More than 10 pills (more than 150mcg/day)
Sufentanil doses 2 | From first day of hospitalization till second day of hospitalization
  Number of pills of sufentanil that the patient has token besides the main treatment. The variable is 2 days after surgery.
  Sufentanil doses 2 is a categorical variable with 4 levels:
  * From 0 to 2 pills (equal or less than 30mcg/day) as level 1.
  * From 2 to 4 pills (from 30mcg/day to 60mcg/day)
  * From 5 to 10 pills (from 75mcg/day to 150 mcg/day)
  * More than 10 pills (more than 150mcg/day)
Sufentanil doses 4 | From second day of hospitalization till fourth day of hospitalization
  Number of pills of sufentanil that the patient has token besides the main treatment. The variable is gathered 4 days after surgery.
  Sufentanil doses 4 is a categorical variable with 4 levels:
  * From 0 to 2 pills (equal or less than 30mcg/day) as level 1.
  * From 2 to 4 pills (from 30mcg/day to 60mcg/day)
  * From 5 to 10 pills (from 75mcg/day to 150 mcg/day)
  * More than 10 pills (more than 150mcg/day)
Sufentanil doses 6 | From fourth day of hospitalization till sixth day of hospitalization
  Number of pills of sufentanil that the patient has token besides the main treatment. The variable is gathered 6 days after surgery.
  Sufentanil doses 6 is a categorical variable with 4 levels:
  * From 0 to 2 pills (equal or less than 30mcg/day) as level 1.
  * From 2 to 4 pills (from 30mcg/day to 60mcg/day)
  * From 5 to 10 pills (from 75mcg/day to 150 mcg/day)
  * More than 10 pills (more than 150mcg/day)
Rescue Methadone | Baseline
  Rescue Methadone is a categorical variable that indicates if the patient required the use of methadone as a secondary treatment besides the main one.
  The variable has 4 levels:
  * No rescue as level 0
  * 5mg/day as level 1
  * From 10mg/day to 15mg/day as level 2
  * More than 15mg/day as level 3
Morphine dosage 1 | From surgery release till first day of hospitalization
  For those cases in which an infusion PCA morphine pump was placed, mean dose 1 day after surgery of the administered morphine.
  Daily morphine dosage is a categorical variable of 4 levels:
  * Less than 30mg/day as level 1
  * From 30mg/day to 60mg/day as level 2
  * From 60mg/day to 150mg/day as level 3
  * More than 150mg/day as level 4
Morphine dosage 2 | From first day of hospitalization till second day of hospitalization
  For those cases in which an infusion PCA morphine pump was placed, mean dose 2 days after surgery of the administered morphine.
  Daily morphine dosage is a categorical variable of 4 levels:
  * Less than 30mg/day as level 1
  * From 30mg/day to 60mg/day as level 2
  * From 60mg/day to 150mg/day as level 3
  * More than 150mg/day as level 4
Morphine dosage 4 | From second day of hospitalization till fourth day of hospitalization
  For those cases in which an infusion PCA morphine pump was placed, mean dose 4 days after surgery of the administered morphine.
  Daily morphine dosage is a categorical variable of 4 levels:
  * Less than 30mg/day as level 1
  * From 30mg/day to 60mg/day as level 2
  * From 60mg/day to 150mg/day as level 3
  * More than 150mg/day as level 4
Morphine dosage 6 | From fourth day of hospitalization till sixth day of hospitalization
  For those cases in which an infusion PCA morphine pump was placed, mean dose 6 days after surgery of the administered morphine.
  Daily morphine dosage is a categorical variable of 4 levels:
  * Less than 30mg/day as level 1
  * From 30mg/day to 60mg/day as level 2
  * From 60mg/day to 150mg/day as level 3
  * More than 150mg/day as level 4
Nausea and vomiting | Baseline
  Nausea and vomiting is a categorical variable that indicates if the patient reported having nausea or vomiting in the control postoperative visits. The variable has 2 states: Yes (1) or No (0).
Intestinal ileus | Baseline
  Intestinal ileus is a categorical variable that indicates if the doctor or nurse reported an intestinal ileus when performing the postoperative control visit. The variable has 2 states: Yes (1) or No (0).
Constipation | Baseline
  Constipation is a categorical variable that indicates if the patient reported having constipation in the control postoperative visits. The variable has 2 states: Yes (1) or No (0).
Anxiolytic rescue agent | Baseline
  The Anxiolytic rescue agent is a categorical variable that indicates if there was a need of applying an axiolytic as a rescue agent besides the main postoperative treatment.
  The variable has 5 levels:
  * Not required as level 0
  * Eventually (1 time per day) as level 1
  * Moderate (2 times per day) as level 2
  * Frequent (3 times per day) as level 3
  * Very Frequently (more than 3 times per day) as level 4
Oral ketamine | Baseline
  Oral ketamine is a categorical variable that indicates if the patient required the use of oral ketamine besides the main postoperative treatment. The variable has 2 states: Yes (1) or No (0).
Chronic opioid and hospital discharge | Up to 6 days
  The Chronic opioid and hospital discharge variable is a categorical variable that resumes the patient state when discharged from the hospital. The variable compares the preoperative opioid dosage with the postoperative dosage prescription.
  The variable has 4 levels:
  * No opioids as level 0
  * Decrease when compared to preoperative (between 20% and 30%) as level 1
  * Same dose when compared to preoperative as level 2
  * More dose when compared to preoperative as level 3

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Rafael Ramirez Paesano, MD, Principal Investigator — Servei d'Anestesiologia Centro Médico Teknon
Locations (1):
- Centro Médico Teknon, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Castori M, Morlino S, Ghibellini G, Celletti C, Camerota F, Grammatico P. Connective tissue, Ehlers-Danlos syndrome(s), and head and cervical pain. Am J Med Genet C Semin Med Genet. 2015 Mar;169C(1):84-96. doi: 10.1002/ajmg.c.31426. Epub 2015 Feb 5. PMID 25655119
- [Background] Henderson FC Sr, Francomano CA, Koby M, Tuchman K, Adcock J, Patel S. Cervical medullary syndrome secondary to craniocervical instability and ventral brainstem compression in hereditary hypermobility connective tissue disorders: 5-year follow-up after craniocervical reduction, fusion, and stabilization. Neurosurg Rev. 2019 Dec;42(4):915-936. doi: 10.1007/s10143-018-01070-4. Epub 2019 Jan 9. PMID 30627832
- [Background] Scheper MC, de Vries JE, Verbunt J, Engelbert RH. Chronic pain in hypermobility syndrome and Ehlers-Danlos syndrome (hypermobility type): it is a challenge. J Pain Res. 2015 Aug 20;8:591-601. doi: 10.2147/JPR.S64251. eCollection 2015. PMID 26316810
- [Background] Lee M, Silverman SM, Hansen H, Patel VB, Manchikanti L. A comprehensive review of opioid-induced hyperalgesia. Pain Physician. 2011 Mar-Apr;14(2):145-61. PMID 21412369
- [Background] Kim DJ, Bengali R, Anderson TA. Opioid-free anesthesia using continuous dexmedetomidine and lidocaine infusions in spine surgery. Korean J Anesthesiol. 2017 Dec;70(6):652-653. doi: 10.4097/kjae.2017.70.6.652. Epub 2017 Apr 21. No abstract available. PMID 29225750
- [Background] Soffin EM, Wetmore DS, Beckman JD, Sheha ED, Vaishnav AS, Albert TJ, Gang CH, Qureshi SA. Opioid-free anesthesia within an enhanced recovery after surgery pathway for minimally invasive lumbar spine surgery: a retrospective matched cohort study. Neurosurg Focus. 2019 Apr 1;46(4):E8. doi: 10.3171/2019.1.FOCUS18645. PMID 30933925
- [Background] Maheshwari K, Avitsian R, Sessler DI, Makarova N, Tanios M, Raza S, Traul D, Rajan S, Manlapaz M, Machado S, Krishnaney A, Machado A, Rosenquist R, Kurz A. Multimodal Analgesic Regimen for Spine Surgery: A Randomized Placebo-controlled Trial. Anesthesiology. 2020 May;132(5):992-1002. doi: 10.1097/ALN.0000000000003143. PMID 32235144
- [Background] Dunn LK, Durieux ME, Nemergut EC. Non-opioid analgesics: Novel approaches to perioperative analgesia for major spine surgery. Best Pract Res Clin Anaesthesiol. 2016 Mar;30(1):79-89. doi: 10.1016/j.bpa.2015.11.002. Epub 2015 Nov 24. PMID 27036605
- [Background] Frauenknecht J, Kirkham KR, Jacot-Guillarmod A, Albrecht E. Analgesic impact of intra-operative opioids vs. opioid-free anaesthesia: a systematic review and meta-analysis. Anaesthesia. 2019 May;74(5):651-662. doi: 10.1111/anae.14582. Epub 2019 Feb 25. PMID 30802933